CLINICAL TRIAL: NCT03054844
Title: Comparison of Two Methods Using Intranasal Lidocaine to Alleviate Discomfort Associated With Administration of Intranasal Midazolam in Children.
Brief Title: PREMIX vs PREMED Intranasal Lidocaine and Midazolam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Pediatrics at CUMC, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAQ6408
Record Dates: First submitted 2017-02-13; First posted 2017-02-16 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Pain
Keywords: Intranasal; Pain; Lidocaine; Midazolam; Emergency department
MeSH Terms: conditions — Pain; Emergencies | interventions — Lidocaine; Midazolam; Premix 730-4

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PREMED (Experimental): Patients will receive 0.25 mL of IN 4% lidocaine (10 mg) in each naris (total of 0.5 mL/20 mg for both nares) preceding adminstration of IN midazolam.
  Interventions: Drug: Lidocaine; Drug: Midazolam
- PREMIX (Experimental): Patients will receive midazolam mixed with 0.5 mL of 4% lidocaine (20 mg).
  Interventions: Drug: Lidocaine and midazolam (PREMIX)

INTERVENTIONS:
Drug: Lidocaine — Lidocaine will be administered before administration of midazolam.
  Other Names: PREMED
  Arms: PREMED
Drug: Lidocaine and midazolam (PREMIX) — Lidocaine will be administered as a mixture with midazolam.
  Other Names: PREMIX
  Arms: PREMIX
Drug: Midazolam — Midazolam will be administered either after lidocaine, or as a mixture with lidocaine.
  Arms: PREMED

SUMMARY:
Intranasal (IN) midazolam is an anxiolytic that is commonly used in the pediatric population for procedural anxiolysis in the emergency department (ED) setting to facilitate painful and distressing procedures, such as laceration repairs. Intranasal midazolam is both effective and safe in children. However, due to the acidic nature of midazolam, there is a burning sensation that is associated with the intranasal administration of midazolam. The use of IN lidocaine has been shown to decrease the pain associated with the administration of IN midazolam and other acidic solutions. The IN lidocaine can be given as a premedication (PREMED), where it is sprayed in the nares first to provide topical anesthesia, and then followed by the administration of the IN midazolam. Lidocaine can also be given concurrently with the IN midazolam (PREMIX), where it is mixed with the midazolam and then the combined mixture administered. Both methods have been shown to be effective in decreasing the pain associated with the intranasal administration of acidic solutions, such as midazolam, although the PREMIX method could have the advantage of requiring less number of sprays, and be tolerated better by children. Although both methods have been shown to work, it is not known if the PREMIX method is non-inferior to the PREMED method for decreasing pain and distress associated with administering IN midazolam. Therefore, the investigators aim to determine if the PREMIX method is non-inferior to the PREMED method of using lidocaine to decrease the pain and distress associated with the administration of IN midazolam in children.

DETAILED DESCRIPTION:
We will enroll 50 children to determine whether the PREMED method is non-inferior to the PREMIX method. We based our sample size on the outcome of pain and distress associated with the administration of IN midazolam, which will be measured using our primary outcome measure of the Observational Scale of Behavioral Distress-Revised (OSBD-R). The OSBD-R is an observational measure of distress that has been well validated in the pediatric population for evaluating painful and distressing procedures, and has been used in children as young as 1 year of age [1,2]. The sample size of 50 patients was determined based on a prestated margin of non-inferiority (delta) of 1.8 (SD 2.25). This value was based on the minimum clinically significant differences used in prior studies of painful procedures in children in the emergency department [3,4,5]. To determine noninferiority using a delta of 1.80 (SD 2.25), with a 1-tailed alpha of 0.025 and power of 80%, we would require 25 patients in each arm, for a total of 50 patients. OSBD-R scores will be determined independently by two blinded trained assessors who will review the videotapes of the study procedures. Interrater reliability of the OSBD-R between the two assessors will evaluated by determining the intraclass correlation coefficient. The period of administration of the midazolam alone in the PREMED group and the period of administration of the midazolam/lidocaine mixture in the PREMIX group are the two phases which will be compared to each other to determine our primary outcome.

Secondary outcome measures of pain and distress associated with IN midazolam administration will include the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS); the Faces-LegsActivity-Crying-Consolability (FLACC) scale; and cry duration. These are all continuous measures that will be analyzed using the independent samples t-test.We will also evaluate parental and provider satisfaction across various domains using a 5-point Likert scale (see attached document for questions to be asked). Responses will be dichotomized into "agree" (i.e. if respondent answers "agree" or "strongly agree") or "disagree" (i.e. if respondent responds "undecided", "disagree", or "strongly disagree") and analyzed using the chi square test.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of ≥ 6 months or ≤ 7 years old
2. Undergoing a laceration repair
3. Treating physician has determined that patient requires intranasal midazolam to facilitate the laceration repair

Exclusion Criteria:

1. Weight < 5 kg
2. Known allergy to Lidocaine or Midazolam
3. Does not speak English or Spanish
4. Nasal injury precluding IN medication delivery
5. Presence of intranasal obstruction (mucous/blood) not easily cleared with suction or nose blowing
6. Baseline motor neurological abnormality (e.g. motor deficit, cerebral palsy)
7. Developmental delay, autism, autism spectrum disorder

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsze DS, Steele DW, Machan JT, Akhlaghi F, Linakis JG. Intranasal ketamine for procedural sedation in pediatric laceration repair: a preliminary report. Pediatr Emerg Care. 2012 Aug;28(8):767-70. doi: 10.1097/PEC.0b013e3182624935. PMID 22858745
- [Background] Tsze DS, Ieni M, Fenster DB, Babineau J, Kriger J, Levin B, Dayan PS. Optimal Volume of Administration of Intranasal Midazolam in Children: A Randomized Clinical Trial. Ann Emerg Med. 2017 May;69(5):600-609. doi: 10.1016/j.annemergmed.2016.08.450. Epub 2016 Nov 4. PMID 27823876
- [Background] Fenster DB, Dayan PS, Babineau J, Aponte-Patel L, Tsze DS. Randomized Trial of Intranasal Fentanyl Versus Intravenous Morphine for Abscess Incision and Drainage. Pediatr Emerg Care. 2018 Sep;34(9):607-612. doi: 10.1097/PEC.0000000000000810. PMID 27387971
- [Background] Godambe SA, Elliot V, Matheny D, Pershad J. Comparison of propofol/fentanyl versus ketamine/midazolam for brief orthopedic procedural sedation in a pediatric emergency department. Pediatrics. 2003 Jul;112(1 Pt 1):116-23. doi: 10.1542/peds.112.1.116. PMID 12837876
- [Background] Lee-Jayaram JJ, Green A, Siembieda J, Gracely EJ, Mull CC, Quintana E, Adirim T. Ketamine/midazolam versus etomidate/fentanyl: procedural sedation for pediatric orthopedic reductions. Pediatr Emerg Care. 2010 Jun;26(6):408-12. doi: 10.1097/PEC.0b013e3181e057cd. PMID 20502386

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PREMED | PREMIX
Started | 28 | 27
Completed | 25 | 26
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Children 6 months to 7 years old with a laceration requiring repair, and intranasal midazolam as determined by their treating physician.
Groups:
- Total: Total of all reporting groups
Arm/Group | PREMED | PREMIX | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2 [2 to 3.5] | 2 [2 to 4] | 2 [2 to 4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 13 | 16 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 16 | 21 | 37
  White | 3 | 1 | 4
  Black | 2 | 2 | 4
  More than one | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Procedural Distress, OSBD-R
Description: The Observational Scale of Behavioral Distress-Revised (OSBD-R) is an observational measure of pain and distress shown to have strong validity in children. The scale is an 8-factor, weighted observational scale used to measure distress associated with medical procedures, which has been validated in children and adults aged 1 to 20 years. The total Observational Scale of Behavioral Distress-Revised score is the sum of the scale scores for each phase, with each phase assigned a score from 0 to 23.5 units on a scale (0=no distress, 23.5=maximum distress), based on the frequency and types of behaviors observed during a predetermined number of 15-second intervals during each phase. There were four phases so the range of scores for the total OSBD-R was 0 to 94 units on a scale, with a higher score indicated a greater degree of distress.
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PREMED | PREMIX
Number analyzed (Participants) | 25 | 26
Units on a scale | 6.4 [5 to 7.8] | 7 [5.2 to 8.9]

2. Secondary Outcome: Procedural Pain
Description: The Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) utilizes six observational factors (cry, facial, verbal, torso, touch, and legs) to evaluate pain in young children and can be used to monitor the effectiveness of interventions for reducing the pain and discomfort of an intervention. This scale rates each behavior numerically, with a score of 4-6 units on a scale representing no pain, and a maximum score of 13 units on a scale representing (most pain perceived).
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PREMED | PREMIX
Number analyzed (Participants) | 25 | 26
Units on a scale | 10.6 [9.7 to 11.4] | 10.5 [9.5 to 11.4]

3. Secondary Outcome: Procedural Distress, FLACC
Description: The Faces, Legs, Activity, Cry, Consolability (FLACC) scale is comprised of five criteria (face, legs, activity, cry, consolability), with a possible score of 0 to 2 units on a scale for each criteria and a possible total score of 0 to 10 units on a scale (0 meaning no pain, 10 meaning most pain).
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PREMED | PREMIX
Number analyzed (Participants) | 25 | 26
Units on a scale | 6.7 [5.3 to 8.1] | 7 [5.4 to 8.6]

4. Secondary Outcome: Procedural Distress, Cry Duration
Description: Cry duration was measured in seconds and defined as the time from onset of crying following administration of an IN medication until the cessation of crying sounds and/or tears. If a patient did not cry, the cry duration was zero
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | PREMED | PREMIX
Number analyzed (Participants) | 25 | 26
seconds | 84 [58 to 109] | 73 [45 to 102]

5. Secondary Outcome: Parental Satisfaction
Description: If my child needed medications to stay calm for a procedure, I would like to use these same medications again.
Time Frame: 1 minute
Measure: Count of Participants; unit: Participants
Arm/Group | PREMED | PREMIX
Number analyzed (Participants) | 25 | 26
Participants | 10 | 12

6. Secondary Outcome: Provider Satisfaction
Description: I would like to use this method of administering intranasal midazolam and lidocaine again in the future
Time Frame: 1 minute
Measure: Count of Participants; unit: Participants
Arm/Group | PREMED | PREMIX
Number analyzed (Participants) | 25 | 26
Participants | 8 | 24

ADVERSE EVENTS:
Time Frame: Course of ED visit, typically between 1-2 hours
Arm/Group | PREMED | PREMIX
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 4/25 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PREMED (N=25) | PREMIX (N=26)
Vomiting (Gastrointestinal disorders) | 3 | 0
Epistaxis (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03054844/Prot_SAP_000.pdf